CLINICAL TRIAL: NCT02577744
Title: Acute Effect of EPAP and Noninvasive Ventilation on Pulmonary Function, Regional Lung Ventilation and Respiratory Mechanics on Patients Submitted Bariatric Surgery Evaluated by Spirometry and Electric Impedance Tomography: A Clinical Trial Controlled Randomized
Brief Title: Acute Effect of EPAP and Noninvasive Ventilation on Pulmonary Function and Lung Regional Ventilation on Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Sóstynis José de Albuquerque Silva, Acute Effect of Epap and Noninvasive Ventilation on Pulmonary Function and Lung Regional Ventilation on Bariatric Surgery, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38032414.3.0000.5208
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Bariatric Surgery; Obesity; Physical Therapy Modalities
Keywords: Electrical Impedance Tomography
MeSH Terms: conditions — Obesity | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Noninvasive Ventilation (Active Comparator): Noninvasive ventilation for 15 minutes with EPAP set at 10 cmH2O and IPAP adjusted to maintain a tidal volume of 6 ml / kg ideal weight.
  Interventions: Other: Noninvasive Ventilation; Other: Expiratory Positive Air Pressure
- Expiratory Positive Air Pressure (Active Comparator): EPAP through facial mask with valve spring load for 15 minutes set at 10 cmH2O.
  Interventions: Other: Noninvasive Ventilation; Other: Expiratory Positive Air Pressure

INTERVENTIONS:
Other: Noninvasive Ventilation — Noninvasive ventilation for 15 minutes with EPAP set at 10 cmH2O and IPAP adjusted to maintain a tidal volume of 6 ml / kg ideal weight.
  Other Names: NIV
Other: Expiratory Positive Air Pressure — EPAP through facial mask with valve spring load for 15 minutes set at 10 cmH2O.
  Other Names: EPAP

SUMMARY:
Obesity is a non-communicable chronic disease of multifactorial, involving biological, historical, ecological, economic, social, cultural and political. Currently, bariatric surgery is considered an effective method of refractory obesity treatment, and only severe obesity effective treatment that leads to reduced long-term weight. It is well documented in the literature regarding the association of abdominal surgery and the incidence of respiratory complications and its main characteristics are: atelectasis, pneumonia, respiratory dysfunction and pleural effusion. All these respiratory complications can be minimized or avoided with the use of a respiratory therapy care protocol, since the pulmonary atelectasis is considered the main cause of complications. An arsenal of resources to physical therapy lung expansion, among these, the application of positive pressure through a valve EPAP (Expiratory positive airway Pressure) and the use of noninvasive ventilation, and aims to prevent and / or improve the complications resulting from postoperative. The electrical impedance tomography (EIT) is an alternate to allow assessment of the respiratory system, without suffering the same interference conditions of patients, such as pain and bed rest. TIE consists of a method that measures passively regional lung ventilation. The aim of this study is to compare the effects of the application of EPAP and NIV on pulmonary ventilation we post bariatric surgery. This is a randomized controlled trial where patients will be divided into two groups: EPAP and NIV and assessed by spirometry, manometer and TIE. The techniques will be applied in the 1st and 2nd postoperative day where they will be evaluated before, during and after the application of the techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bariatric surgery, of both sexes and aged between 20 and 50 years.

Exclusion Criteria:

* severe lung disease;
* patients with congestive heart failure (NYHA Class III or IV);
* coronary artery disease;
* presented hemodynamic instability (MAP <60 mmHg) or arrhythmias during the performance of techniques, plus any contraindications to perform the BS techniques, EPAP and NIV to consider: Trauma / facial injury that prevents the attachment of the mask, extreme anxiety, hypotension and lack of patient cooperation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Regional Pulmonary Ventilation | six months
  Assessment of regional ventilation through the variables of electrical impedance tomography , Delta Z (impedance variation) in the anterior and posterior region, and right and left lung.

SECONDARY OUTCOMES:
Effects of bariatric surgery on respiratory muscle strength | Six months
  Assessment of maximum inspiratory pressure by manometer before and after bariatric surgery .
Patient perception of evaluation and assessing the quality of postoperative recovery | Six months
  Evaluation by applying the Global Quality of recovery -40 questionnaire (QoR -40) at 24 and 48 hours after the surgical procedure.
Effects of bariatric surgery on lung function | Six months
  Evaluation by spirometry, considering the variables, CV, FEV1, FVC, PEF, FEV1/FVC, FEF 25-75 %.
Adverse effects of technical and EPAP NIV | Six months
  Through evaluation of open questions about the occurrence of adverse effects during the technique, such as headache, nausea, dizziness, discomfort, nausea and vomiting.
Therapeutic effect time of the EPAP and NIV | six months
  Quantify the therapeutic effect of time of the technical EPAP and NIV by analyzing the variables of the impedance electrical tomography , Average electrical impedance at the end of expiration (MIEFE) and monitoring this baseline during the post technique period at times 5 and 30 minutes post intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas, Recife, Pernambuco, Brazil